CLINICAL TRIAL: NCT05306301
Title: Combination of Ponatinib Plus Chemotherapy As Frontline Treatment For Patients With BCR/ABL1-Like Acute Lymphoblastic Leukemia (BCR/ABL1-Like ALL)
Brief Title: Ponatinib Plus Chemotherapy in Acute Lymphoblastic Leukemia Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL2922
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Chemotherapy; Leukemia, Acute Lymphoblastic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients With BCR/ABL1-Like Acute Lymphoblastic Leukemia (Experimental): In the run-in phase, patients will receive a dosage of 15 mg of ICLUSIG (ponatinib). If there are no toxicities observed, 30 mg of ponatinib will be administered in the remaining patients. MRD of patients will be evaluated on weeks 4, 10, 16, and 22. If a donor is available, MRD-positive patients will proceed to an allogeneic transplant after cycle 3. If there is no donor available, they'll continue treatment with 5 additional consolidation/reinduction blocks, followed by 24 28-day cycles of maintenance.
  Induction/consolidation cycles are administered at 28 (cycles 1-2) and 21(cycles 2-8) day intervals.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib is a novel, synthetic, orally-active TKI discovered using a computational and structure based drug design approach. Ponatinib was specifically designed to inhibit all clinically relevant variants of BCR-ABL1, including the T315I mutant (15-17). In vitro assays have demonstrated that Ponatinib potently inhibits the kinase enzymatic activity of the T315I ABL kinase domain, as well as that of the native (unmutated) enzyme. In leukemia cell lines expressing these BCR-ABL1 variants, Ponatinib potently inhibited BCR-ABL1 signaling, leading to the reduction of cellular proliferation and induction of apoptosis. Ponatinib also inhibits the proliferation of cell lines expressing other major clinically-observed Imatinib-resistant mutants of BCR-ABL1.

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most frequent cancer in children, decreases in adolescence and adulthood, and a second peak can be recorded starting from the 6th decade of life. While the outcome in children is excellent, in the adolescent/adult population, the prognosis, though improved over the decades, it is still unsatisfactory and novel biologically-driven approaches are urgently needed. In this setting, thanks to the introduction of genome wide technologies, it was possible to recognize specific subset of ALL. Among those, the BCR/ABL1-like ALL are of extreme importance, since they are characterized by an unfavourable outcome and, on the other hand, can benefit of a targeted treatment, in particular with the pan-tyrosine kinase inhibitor ponatinib.

The primary objective is to evaluate the clinical response - in terms of MRD negativity - in patients with a BCR/ABL1-like profile, according to the BCR/ABL1-like predictor tool, treated with Ponatinib in combination with chemotherapy.

DETAILED DESCRIPTION:
This is an interventional, phase II study, foreseeing a run-in phase for adult BCR/ABL1-like ALL patients. Thirty-two newly-diagnosed B-lineage ALL cases with a BCR/ABL1-like profile will be treated (≥18 years old, up to the age of 65 years). This implies that about 100-120 B-lineage ALL patients negative at the conventional molecular screening (BCR/ABL1, ALL1/AF4, E2A/PBX1) will undergo the recently reported "BCR/ABL1 predictor" (13). The estimated timing for both the conventional and the BCR/ABL1-like screening is within the steroid pre-phase (7 days). After a steroid pre-treatment phase (prednisone: 60 mg/m2/day, day -6 up to day 0), that can occurr before enrollment during the screening period, patients who prove BCR/ABL1-like will be treated with Ponatinib in combination with a pediatric-inspired and minimal residual disease (MRD)-driven treatment scheme - as in the previous GIMEMA LAL1913 protocol (EudraCT number 2009-016075-30) -, for the first 2 cycles (C1 and C2). In order to avoid toxicity, namely thrombotic, pancreatic and hepatic events, Asparaginase will be omitted from this scheme. As for the run-in phase, patients will receive ponatinib at the dosage of 15 mg. If no relevant toxicities are observed (i.e. 2 distinct patients developing a Grade IV non hematologic toxicity related to ponatinib within the first cycle of induction, 28 days), Ponatinib will be administered at the dose of 30 mg in the remaining patients. MRD will be evaluated at week 4, 10, 16, and 22. If a donor is available (MUD and haploidentical donors allowed, HLA typing carried out as soon as possible), MRD-positive patients will proceed to an allogeneic transplant after cycle 3; otherwise, if no donor is available, they will continue treatment with 5 additional consolidation/reinduction blocks, followed by 24 28-day cycles of maintenance, as detaield in the treatment scheme. If beneficial for the patients, ponatinib will be provided until disease progression. CNS prophylaxis will be carried out throughout the course of treatment with 12 medicated rachicenteses (Methotrexate 12.5 mg, Aracytin 50 mg, Urbason 20 mg).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* De novo Ph+-like ALL, as defined by the BCR/ABL1-like predictor (13).
* WHO score ≤2.
* Adequate liver function, as defined by the following criteria: total serum bilirubin ≤1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, alanine aminotransferase (ALT) ≤2.5 × ULN or ≤2.5 x ULN or leukemia related.
* Adequate pancreatic function as defined by serum lipase and amylase ≤1.5 × ULN or leukemia related.
* No history of dyslipidemia, thrombotic events or cardiac disease.
* For females of childbearing potential, a negative pregnancy test must be documented.
* Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from enrollment through 12 months after the end of treatment.
* Signed informed consent, according to ICH/EU/GCP and national regulation.

Exclusion Criteria:

* WHO performance status >2.
* Active HBV or HCV hepatitis, or AST/ALT > 2.5 x ULN and bilirubin > 1.5 x ULN.
* History of acute pancreatitis within 1 year of study or history of chronic pancreatitis.
* History of alcohol abuse.
* Ongoing or active infections.
* Uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL).
* Clinically significant, uncontrolled or active cardiovascular disease, specifically including, but not restricted to:
* Any history of myocardial infarction, stroke, or revascularization, unstable angina or transient ischemic attack within 6 months prior to enrollment,
* Congestive heart failure within 6 months prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards,
* History of clinically significant (as determined by the treating physician) atrial arrhythmia,
* Any history of ventricular arrhythmia,
* Any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism.
* Uncontrolled hypertension (diastolic blood pressure >90 mm Hg; systolic >140 mm Hg). Patients with hypertension should be under treatment on study entry to effect blood pressure control.
* Taking medications that are known to be associated with torsades de pointes.
* Taking any medications or herbal supplements that are known to be strong inhibitors of CYP3A4 within at least 14 days before the first dose of ponatinib.
* Creatinine levels > 2.5mg/dl or glomerular filtration rate (GFR) < 20 ml/min or proteinuria >3.5 g/day.
* Gastrointestinal (GI) function impairment, or a GI disease that may significantly alter the absorption of study drugs.
* Patients who are currently receiving treatment with any of the medications with potential to prolong QT interval (listed in Appendix F) if the medications cannot be either discontinued or switched to a different medication prior to starting study drug.
* Patients who have received any investigational drug ≤ 4 weeks.
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who are pregnant or breast feeding and adults of reproductive potential not employing an effective method of birth control (women of childbearing potential must have a negative serum pregnancy test within 48 hrs. prior to administration of Ponatinib). Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ two effective reliable methods of birth control throughout the study and for up to 12 months following discontinuation of study drugs.
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients unwilling or unable to comply with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
MRD Negativity Rate after 3 cycles (TP2) in patients with BCR/ABL1-like ALL treated with a Ponatinib plus chemotherapy approach | 3 months
  The primary outcome is to evaluate the clinical response - in terms of MRD negativity - in patients with a BCR/ABL1-like profile, according to the BCR/ABL1-like predictor tool, treated with Ponatinib in combination with chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Chiaretti, Principal Investigator — Ematologia - Policlinico Umberto I di Roma
Locations (24):
- Italy (24):
  - Ematologia con Unità di Trapianto, Avellino, AV
  - Ematologia Presidio Ospedaliero Tortora, Pagani, SA
  - Ematologia ASST Papa Giovanni XXIII, Bergamo
  - Ematologia AOU S.ORSOLA-MALPIGHI, Bologna
  - Ematologia ASST Spedali Civili, Brescia
  - Ematologia AOU Policlinico Vittorio Emanuele-Ferrarotto, Catania
  - Ematologia AOU Careggi, Florence
  - Ematologia Ospedale V.Fazzi, Lecce
  - Ematologia Ospedale dell'Angelo, Mestre
  - Ematologia Ospedale Maggiore Policlinico, Milan
  - Ematologia AOU Federico II, Napoli
  - Ematologia AOU Maggiore della Carità, Novara
  - Ematologia AO Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Ematologia Fondazione Policlinico San Matteo, Pavia
  - Ematologia Presidio Ospedaliero Spirito Santo, Pescara
  - Ematologi Presidio Ospedaliero Guglielmo da Saliceto, Piacenza
  - Ematologia Presidio Ospedaliero Infermi, Rimini
  - Dipartimento di Medicina Traslazionale e di Precisione - Ematologia, Roma
  - Ematologia AOU Policlinico Tor Vergata, Roma
  - Ematologia Policlinico A.Gemelli, Roma
  - Ematologia AOU Senese, Siena
  - Ematologia Ospedale Mauriziano, Torino
  - Ematologia Ospedale S.Giovanni Battista Molinette, Torino
  - Ematologia Policlinico G.B. Rossi, Verona